CLINICAL TRIAL: NCT01574755
Title: Long Term Outcome of Argon Plasma Coagulation of Cervical Heterotopic Gastric Mucosa as an Alternative Treatment for Globus Sensations
Acronym: ACHAT FU
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: ACHAT-FU-1
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Globus Sensations in the Throat
Keywords: gastric inlet patches; argon plasma coagulation; globus sensations
MeSH Terms: conditions — Globus Sensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — biopsy of gastric inlet patches
Oversight: Data Monitoring Committee: No

SUMMARY:
APC of gastric inlet patches is successful for the treatment of globus sensations in the throat (Bajbouj et al Gastroenterology 2009; 137:440-4). There is no data for long term efficiency of this treatment. To measure long term efficacy all patients treated with this therapy in our clinic were followed up with complaint-evaluation sheets and endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* former APC therapy of gastric inlet patches as treatment for globus sensations
* at least 6 month since last APC therapy

Exclusion Criteria:

* patients with reduced general condition
* malignancy of the upper gastrointestinal tract
* patients older than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient clinic of a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change of globus complaint score | retrospectively assessed: before APC therapy and at the date of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Departmet for Internal Medicine and Gastroenterology, Technical University Munich, Germany; Alexander Meining, Professor, Study Chair — Department for Internal Medicine and Gastroenterology, Technical University Munich, Germany; Monther Bajbouj, Assistent Professor, Study Director — Department for Internal Medicine and Gastroenterology, Technical University Munich, Germany